CLINICAL TRIAL: NCT03713736
Title: Papillomavirus Load in Rheumatic Inflammatory Diseases
Acronym: PAPLOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0539
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-06

CONDITIONS: Spondyloarthritis; Rhumatoid Arthisis
Keywords: HPV infection; Spondyloarthritis; Rhumatoid Arthritis; Cervical smear; cervical cancer screening
MeSH Terms: conditions — Spondylarthritis; Papillomavirus Infections | interventions — Vaginal Smears; Human Papillomavirus DNA Tests; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female patients with spondyloarthritis or rheumatoid arthritis (Other): Female patients (18 to 65 years old) with spondyloarthritis or rheumatoid arthritis will undergo HPV screening and a have a close gynecologic follow-up.
  Interventions: Diagnostic Test: Cervical smear; Diagnostic Test: Pregnancy test; Behavioral: Sexual activity questionnary

INTERVENTIONS:
Diagnostic Test: Cervical smear — Cervical smear will be obtained using an Ayre spatula and a cervical brush (Cervex-Brush®). HPV test will be performed using the CLART® HPV2 kit (Genomica).This kit enables the detection of 35 genotypes: HPV6, 11, 16, 18, 26, 31, 33, 35, 39, 40, 42, 43,44, 45, 51, 52, 53, 54, 56, 58, 59, 61, 62, 66, 68, 70, 71, 72, 73, 81, 82, 83, 84, 85 et 89.
  Other Names: HPV test
Diagnostic Test: Pregnancy test — Urinary pregnancy test
Behavioral: Sexual activity questionnary — Sexual activity questionnary

SUMMARY:
Rheumatoid arthritis (RA) and spondyloarthritis (SpA) are the two most common chronic inflammatory rheumatism, with a prevalence in the French population of 0.3% and 0.4%, according to the criteria European League Against Rheumatism / American College of Rheumatology (EULAR / ACR) 2010 and Assessemnt of SpondyloArthritis International Society (ASAS) 2009 respectively. In patients whose pathology is resistant to first-line treatment, such as methotrexate for rheumatoid arthritis and peripheral spondyloarthritis, or non-steroidal anti-inflammatory drugs for axial spondyloarthritis, the treatment is based on biotherapies, such as anti-inflammatory drugs. -TNF, to obtain effective control of the disease and prevent joint damage.

Human papillomavirus (HPV) infection, the leading risk factor for cervical carcinoma, is the most common sexually transmitted infection (STI) with a particularly high prevalence among young women.

In addition, anti-TNF, used in the treatment of RA and SpA, and anti-IL6 receptor, used in that of RA, could have opposite effects on HPV-dependent oncogenesis.

Thus, patients with RA or SpA may have a higher risk than the general population of progression to cervical cytological abnormalities. Evaluation of the chronic carriage of HPV would then be a useful tool in the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Woman between 18 and 65 years old
* Patient with rheumatoid arthritis as defined in 2010 ACR/EULAR criteria or with spondyloarthritis as defined in 2009 ASAS criteria
* Patient able to understand the objectives of the study and give documented informed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or breastfeeding patient
* Patient with a history of cervical cancer
* Patient under juridical protection
* Patient unable to provide informed consent due to linguistic or psychic impairment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 385 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-01-09 (Estimated); Study Completion 2024-01-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of papillomavirus chronic load in women with rheumatic inflammatory diseases (rheumatoid arthritis and spondyloarthritis), compared to the prevalence in general population | At the end of the 24 months follow-up.
  Papillomavirus chronic load is defined as a positive HPV test at the end of the study combined with at least 3 positive HPV tests during the 24 months follow-up.

SECONDARY OUTCOMES:
To determine the prevalence of HPV infections, whatever the type of HPV | At enrollment
  Number of patients with a positive HPV test at enrollment
To determine the incidence of HPV infection in women with a negative HPV test at enrollment. | At 24 months.
  Number of patients with a negative HPV test at enrollment and having at least one positive HPV test during the 24 months follow-up
To determine the clearance of HPV with women with appositive HPV test at enrollment | At 24 months
  Number of patients with a positive HPV test at enrollment and having a negative HPV test at the end of the study.
To evaluate the incidence of cytological abnormalities in women with normal cytology at enrollment according to HPV chronic load and type. | At 24 months.
  Number of patients with low-grade and high-grade cytological abnormalities during follow-up among those who had normal cytology at enrollment.
To determine the evolution (regression, persistence or invasion) of cytological abnormalities in women with abnormal cytology at enrollment and according to HPV chronic load and type. | At 24 months.
  Number of patients ,with normal cytology at enrollment, whose cervical smear indicates a regression in cytological abnormalities or a persistence of cytological abnormalities or a development of abnormalities into cervical cancer or dysplasia, during the 24 months follow-up.
To determine the number of conization according to HPV chronic load and type. | At 24 months.
  Number of conization

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne COURY-LUCAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Department of obstetrics, Femme Mère Enfant Hospital, Lyon, France, Bron
  - Hopital Edouard Herriot - service de rhumatologie, Lyon
  - Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No